CLINICAL TRIAL: NCT03261583
Title: Impact of Preoperative Martial Deficiency on the Level of Blood Transfusion in Programmed Cardiac Surgery (CARMATS)
Brief Title: Impact of Preoperative Martial Deficiency on the Level of Blood Transfusion in Programmed Cardiac Surgery
Acronym: CARMATS
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC16_3051_CARMATS
Record Dates: First submitted 2017-08-23; First posted 2017-08-25 (Actual); Last update posted 2018-09-18 (Actual); Status verified 2018-09

CONDITIONS: Thoracic Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Thoracic Surgery: Observational study. It is only a matter of collecting clinical data.
  Interventions: Other: Thoracis Surgery - Common care

INTERVENTIONS:
Other: Thoracis Surgery - Common care — Observational study. It is only a matter of collecting clinical data.

SUMMARY:
Observational study.

DETAILED DESCRIPTION:
Blood transfusion is expensive, and has medical and safety consequences for patients who benefit from it. In cardiac surgery, the data concerning the level of perioperative transfusion are very heterogeneous from one center to another. In a large US cohort study of 798 cardiac surgery centers and 102,470 patients undergoing coronary artery bypass surgery, the rate of blood transfusion varies from 8 to 93% depending on the center. It would appear that the largest and most experienced centers have a blood transfusion rate of around 60%.

In addition to its beneficial role in reducing mortality induced by deep or poorly tolerated anemia, current data from the literature also raise morbidity and mortality related to blood transfusion. Murphy et al. Have shown, in an English cohort of cardiac surgery, that transfusion of CGR was correlated with the occurrence of postoperative infections and ischemic events, as well as early and late excess mortality. These effects appear as early as the first transfused red blood cell, which is confirmed by a prospective Brazilian study with a hazard ratio of death occurrence of 1.2 for each RBC transfused after cardiac surgery.

Preoperative anemia is found in 25% of patients in programmed cardiac surgery and its etiologies are varied. Iron deficiency appears to be at the forefront, especially in coronary patients for whom studies report up to 48% iron deficiency anemia. It may also be vitamin B12 deficiency or folate, chronic pathologies such as renal insufficiency, or any other common cause of anemia.

According to the latest European recommendations, iron deficiency should be defined as <100 ng / mL ferritin or <300 ng / mL ferritin combined with a transferrin saturation <20%.

In cardiac surgery, iron deficiency affects 37% of preoperative patients and is associated with more frequent preoperative and postoperative anemia. It is an independent risk factor for postoperative blood transfusion, even in the absence of preoperatively associated anemia It is currently recommended to seek iron deficiency preoperatively during the discovery of any microcytic anemia and to achieve iron substitution if found. And also to seek supplemental iron deficiency in all patients with cardiac insufficiency.

ELIGIBILITY:
Inclusion Criteria:

All adult patients programmed for cardiac surgery in the cardiothoracic surgery departments of Rennes, Poitiers, and Brest.

Exclusion Criteria:

* Children <18 years;
* Procedures for endovascular surgery;
* Vascular surgery other than ascending aorta and lacrosse;
* Non-cardiac thoracic surgery;
* Persons of full age who are subject to legal protection (safeguard of justice, curatorship, guardianship), persons deprived of their liberty.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients programmed for cardiac surgery
Sampling Method: Non-Probability Sample
Enrollment: 444 (Actual)
Dates: Start 2016-11-14 (Actual); Primary Completion 2018-01-15 (Actual); Study Completion 2018-01-15 (Actual)

PRIMARY OUTCOMES:
Incidence of patients with iron deficiency | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Baptiste Gaudriot, Principal Investigator — CHU Rennes
Locations (2):
- France (2):
  - Brest University Hospital, Brest
  - Rennes University Hospital, Rennes